CLINICAL TRIAL: NCT01240408
Title: E7080 Food Effect Study in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: E7080-A001-003
Record Dates: First submitted 2010-11-11; First posted 2010-11-15 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2013-11

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment group 1 (Experimental): 10 mg lenvatinib (1x10 mg lenvatinib capsule) with food
  Interventions: Drug: HOPE
- Treatment group 2 (Experimental): 10 mg lenvatinib (1x10 mg lenvatinib capsule) without food
  Interventions: Drug: HOPE

INTERVENTIONS:
Drug: HOPE — 10 mg lenvatinib (1x10 mg lenvatinib capsule) with food
  Other Names: E7080
  Arms: Treatment group 1
Drug: HOPE — 10 mg lenvatinib (1x10 mg lenvatinib capsule) without food
  Other Names: E7080
  Arms: Treatment group 2

SUMMARY:
This will be a randomized, single-dose, open-label, two-period crossover study in 16 healthy subjects. The study will consist of two phases: Pre-randomization and Randomization. The Pre-randomization phase will have two periods: Screening and Baseline. In the Randomization Phase, subjects will be randomized to one of two possible treatment sequences (fed/fasted and fasted/fed). In each period, subjects will receive a single capsule containing 10 mg lenvatinib either with or without a standard breakfast. There will be a 2-week washout between treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, male or female subjects age greater than or equal to 18 years and less than or equal to 55 years old;
2. Body mass index (BMI) greater than 18 and less than or equal to 32 kg/m2 at Screening;
3. All females must have a negative serum B-human chorionic gonadotropin (B-hCG) test result or negative urine pregnancy test results at Screening and Baseline. Females of child-bearing potential must agree to use a medically acceptable method of contraception (eg, abstinence, an intrauterine device, a double-barrier method such as condom + spermicide or condom + diaphragm with spermicide, a contraceptive implant, an oral contraceptive or have a vasectomised partner) throughout the entire study period and for 30 days after study drug discontinuation. The only subjects who will be exempt from this requirement are postmenopausal women (defined as greater than age 50 and with at least 12 months of amenorrhea) or subjects who have been sterilized surgically or who are otherwise proven sterile (eg, bilateral tubal ligation with surgery at least 6 months prior to dosing, hysterectomy, or bilateral oophorectomy with surgery at least 2 months prior to dosing). All women who are of reproductive potential and who are using hormonal contraceptives must have been on a stable dose of the same hormonal contraceptive product for at least 12 weeks prior to dosing and must continue to use the same contraceptive during the study and for 30 days after study drug discontinuation;
4. Male subjects who are partners of women of childbearing potential must use, or their partners must use a highly effective method of contraception (eg, condom + spermicide, condom + diaphragm with spermicide, intrauterine device (IUD) starting for at least one menstrual cycle prior to starting study drug(s) and throughout the entire study period and for 30 days (longer if appropriate) after the last dose of study drug). Those with partners using hormonal contraceptives must also be using an additional approved method of contraception (as described previously);
5. Provide written informed consent;
6. Are willing and able to comply with all aspects of the protocol.

Exclusion Criteria:

1. Evidence of clinically significant cardiovascular, hepatic, gastrointestinal, renal, respiratory, endocrine, hematological, neurological, or psychiatric disease or abnormalities or a known history of any gastrointestinal surgery that could impact the pharmacokinetics of study drug;
2. A clinically significant illness within 8 weeks or a clinically significant infection within 4 weeks, of dosing;
3. Evidence of organ dysfunction or any clinically significant deviation from normal in their medical history;
4. History of clinically significant drug or food allergies or presently experiencing seasonal allergies;
5. Evidence of clinically significant deviation from normal in physical examination, vital signs, electrocardiograms (ECG) or clinical laboratory determinations at Screening or Baseline;
6. Clinically significant ECG abnormality including a marked baseline prolongation of QT/QTc interval (eg repeated demonstration of a QTc interval greater than 500 msec), or a family history of prolonged QTc syndrome or sudden death;
7. History of drug or alcohol misuse within 6 months prior to Screening, or who have a positive urine drug test at Screening or Baseline;
8. Positive result for Hepatitis B surface antigen (HBsAg) or Hepatitis C antibody (HCV) screen, or a positive syphilis screen;
9. Diagnosed with acquired immune deficiency syndrome (AIDS), or test positive for human immunodeficiency virus (HIV);
10. Participated in another clinical trial less than 4 weeks prior to dosing or who are currently enrolled in another clinical trial;
11. Consumed caffeinated beverages or food within 72 hours prior to dosing;
12. Consumed grapefruit or grapefruit containing beverages or food within 72 hours prior to dosing;
13. Experienced a weight loss or gain of greater than 10% within 4 weeks of dosing;
14. Engaged in heavy exercise (greater than or equal to 1 hour/day 5 times/week) less than 2 weeks prior to Baseline (eg, marathon runners, weight lifters, etc.);
15. Received blood products within 4 weeks, or donated blood within 8 weeks, or donated plasma within 1 week, of dosing;
16. Hemoglobin level less than 12.0 g/dL;
17. Used prescription drugs within 2 weeks prior to screening;
18. Taken over-the-counter (OTC) medications within 2 weeks prior to dosing;
19. Any condition that would make him/her in the opinion of the Investigator or Sponsor, unsuitable for the study or who, in the opinion of the Investigator, is not likely to complete the study for any reason;
20. Inability to tolerate venepuncture and/or venous access;
21. History of depression, deliberate self harm or suicidal ideation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2010-07; Primary Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
To determine the effect of food on the bioavailability of lenvatinib. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Eisai Inc.
Locations (1):
- Charles River Clinical Studies, NW, Tacoma, Washington, United States